CLINICAL TRIAL: NCT03519113
Title: Dose Selection(Step 1), Non-inferiority(Step 2), Phase II/III Clinical Trials to Evaluated the Efficacy and Safety of Hepatitis B Virus-associated Liver Transplant Patients by Intravenously Injecting GC1102
Brief Title: HBV-associated Liver Transplant(LT) Patients by IV Injecting GC1102
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GC1102_P2b/3
Record Dates: First submitted 2018-03-20; First posted 2018-05-08 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2019-10

CONDITIONS: Hepatitis B Infection
Keywords: HBV-related liver transplantation; Hepatitis B immunoglobulin
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test group 1 (Experimental): GC1102 80,000 IU
  Interventions: Biological: GC1102 80,000 IU
- Test group 2 (Experimental): GC1102 100,000 IU
  Interventions: Biological: GC1102 100,000 IU
- Control group (Active Comparator): I.V HBIG
  Interventions: Biological: I.V HBIG

INTERVENTIONS:
Biological: GC1102 80,000 IU — recombinant human hepatitis B immunoglobulin
  Arms: Test group 1
Biological: GC1102 100,000 IU — recombinant human hepatitis B immunoglobulin
  Arms: Test group 2
Biological: I.V HBIG — human anti-hepatitis B Immunoglobulin
  Arms: Control group

SUMMARY:
This is a clinical study for GC1102 to demonstrate preventing the recurrence of hepatitis B virus (HBV) infection following liver transplantation and a dose-finding study to determine its optional dose.

DETAILED DESCRIPTION:
GC1102 is a new recombinant hepatitis B immunoglobulin (HBIG) from Chinese Hamster Ovary (CHO) cells. It is a monoclonal antibody and has high affinity and avidity to hepatitis B surface antigen and several advantages compared to HBIG derived from blood plasma of human donors. Volunteers will participate in the study, receive 24-week treatment with 80,000/100,000 IU of GC1102 or I.V HBIG and be followed up till 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who was informed of, and fully understood, all aspects of the study and has provided voluntary written consent for participation in the study
2. Subject aged over 19 years at the time of consent provided
3. Subject with planned liver transplantation due to HBV-related end-stage liver disease such as cirrhosis, liver cancer and fulminant hepatic failure
4. Subject with HBsAg(+)

Exclusion Criteria:

1. Subject with planned reoperation following liver transplantation
2. Subject with hemophilia
3. Subject with a history of venous or arterial thrombosis
4. Subject with HAV, HCV or HIV infection
5. Subject with immunodeficiency or immunosuppression due to whole body steroids before liver transplantation
6. Subject with hemolytic or blood loss anemia
7. Subject with IgA deficiency
8. Subject with a history of malignant tumor within the last 5 years, excluding primary liver cancer
9. Subject with moderate to severe kidney disease (serum creatinine > 20mg/dL or anuria, kidney failure or dialysis)
10. Subject with a history of transient ischemic attack(TIA), myocardial infarction(MI), unstable angina, cerebral infarction, cerebral hemorrhage, percutaneous transluminal angioplasty(PTA) or coronary artery bypass graft(CABG) within the last 6 months prior to the screening
11. Subject with severe heart failure(NYHA class III~IV), arrythmia requiring treatment
12. Subject with known hypersensitivity (anaphylaxis) to any component of the study drug
13. Subject who had received other immunoglobulin product within the last 3 months prior to the study entry
14. Subject who had received live parenteral vaccine (MMR, Cholera and Varicella) within the last 3 months prior to the study entry
15. Subject who had received estrogen or hormone alternative medicine
16. Pregnant or breast-feeding women
17. Woman of childbearing potential with positive pregnancy test confirmed by serum beta-human chorionic gonadotropin(B-HCG) test within 28 days prior to dosing by urine pregnancy or Subject who refused to use a reliable method of contraception
18. Alcohol or drug abuse within 6 months
19. Subject who has participated in any other clinical trial within 30 days
20. Subject who has any clinically meaningful disease investigator's judgement to prevent participating in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2018-03-29 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevention Failure rate of HBV | 28weeks
  Seroconversion rate of HBsAg or HBeAg, anti-HBs < 500 IU/L

SECONDARY OUTCOMES:
Recurrence rate of HBV | 28weeks
  Seroconversion rate of HBsAg or HBeAg
Prophylactic failure rate of HBV | 28weeks
  Seroconversion rate of HBsAg or HBeAg, anti-HBs < 500 IU/L
Recurrence duration | 28weeks
  Seroconversion time of HBsAg or HBeAg
Overall survival rate | 1 year
  survival rate during 1 year
Geometric mean titer of HBV DNA | 1 year
  Geometric mean titer(GMT) of HBV DNA
Change of anti-HBe | 1 year
  anti-hepatitis B e(HBe)

OTHER OUTCOMES:
Pharmacokinetic(PK) parameters | 1 year
  serum drug titer
Area under curve(AUC) | 1 year
  area under the baseline corrected serum titer versus time curve from time 0 to time of the last measureable titer
clearance(CL) | 1 year
  clearance
Vdss | 1 year
  volume of distribution
Vdss/CL | 1 year
  effective half-life
Adverse events | 1 year
  Adverse events occured during clinical trials
Clinical abnormalities | 1 year
  Clinical laboratory test

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Gyu Lee, Ph.D, Principal Investigator — Seoul Asan Medical Center
Locations (1):
- Seoul Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No